CLINICAL TRIAL: NCT01515319
Title: A Randomised, Placebo Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Y242 in Adult Subjects
Brief Title: Safety and Pharmacokinetic Study of Y242 in Adult Subjects
Acronym: Y242-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: QLON/2011/Y242-01; 2011-003549-17 (EudraCT Number)
Record Dates: First submitted 2011-12-22; First posted 2012-01-24 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Obesity
Keywords: Obesity; Peptide YY; Food intake; Safety; Pharmacokinetics
MeSH Terms: conditions — Obesity | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Part A was a single blind, randomised, placebo controlled, single ascending dose (SAD) study.
  Part B was a double blind, randomised, placebo controlled, multiple ascending dose (MAD) study
Who Masked: Participant, Investigator
Masking Description: Part A: Treatments were administered single-blind; subjects were blinded with regard to treatment and clinical staff remained blinded with regard to treatment until the Safety Committee meeting. Part B was double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- 2mg Y242 (Part A) (Experimental): Y242 single dose, subcutaneous
  Interventions: Drug: Y242
- 7.5mg Y242 (Part A) (Experimental): Y242 single dose, subcutaneous
  Interventions: Drug: Y242
- 15mg Y242 (Part A) (Experimental): Y242 single dose, subcutaneous
  Interventions: Drug: Y242
- 30mg Y242 (Part A) (Experimental): Y242 single dose, subcutaneous
  Interventions: Drug: Y242
- 60mg Y242 (Part A) (Experimental): Y242 single dose, subcutaneous
  Interventions: Drug: Y242
- 90mg Y242 (Part A) (Experimental): Y242 single dose, subcutaneous
  Interventions: Drug: Y242
- Placebo - Part A (Placebo Comparator): 0.9% saline
  Interventions: Drug: 0.9% saline
- 60mg Y242 (Part B1) (Experimental): Y242 single subcutaneous dose, administered once a week for 5 weeks
  Interventions: Drug: Y242
- 90mg Y242 (Part B2-B4) (Experimental): Y242 single subcutaneous dose, administered once a week for 5 weeks
  Interventions: Drug: Y242
- Placebo - Part B (Placebo Comparator): 0.9% saline
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Y242 — Single ascending dose: subcutaneous injection of 2, 7.5, 15, 30, 60 and 90 mg Y242 (Part A); Multiple ascending dose: Y242 single subcutaneous dose, administered once a week for 5 weeks (Part B)
  Arms: 15mg Y242 (Part A); 2mg Y242 (Part A); 30mg Y242 (Part A); 60mg Y242 (Part A); 60mg Y242 (Part B1); 7.5mg Y242 (Part A); 90mg Y242 (Part A); 90mg Y242 (Part B2-B4)
Drug: 0.9% saline — Identical volume to that of Y242
  Arms: Placebo - Part A; Placebo - Part B

SUMMARY:
Obesity causes 600 premature deaths per week in the UK and existing treatments are not effective. When humans eat, the bowels naturally secrete chemicals into the bloodstream which make people feel full and which stop eating. One of these chemicals is known as Peptide YY (PYY). The investigators have previously shown that injections of PYY reduce appetite and food intake in human volunteers. The investigators have now developed a very similar chemical, Y242, as a treatment for obesity. Y242 has been tested in animals and has been shown to be safe, to reduce their appetite, and to last for much longer than PYY itself. This study will test Y242 to ensure that it is well tolerated in humans, and to see how long it lasts in the blood stream after being injected under the skin. It will also look for any effects on appetite.

DETAILED DESCRIPTION:
Obesity causes 600 premature deaths per week in the UK and existing treatments are less than ideal. Intravenous infusion of a hormone called PYY reduces food intake but its effects only last for a few hours and it can cause nausea. Y242 is a longacting analogue of PYY. Given subcutaneously in rodents, it has a profile of action of at least 72 hours and strongly inhibits food intake. It causes weight loss without behavioural effects. With MRC funding, Y242 has passed Good Laboratory Practice toxicology testing and the present proposal is a first in human study to investigate its safety, tolerability and pharmacokinetics in overweight but otherwise healthy men.

The study is a combined single ascending dose (part A) and multiple ascending dose (part B) Phase 1 investigation. The primary objective is to investigate safety and tolerability. The secondary objective is to assess Y242's pharmacokinetic (PK) profile. Possible effects on food consumption will be explored. For part A up to 48 subjects are planned, with up to 40 subjects for part B. In each part subjects are divided into groups, each of which is dosed with the same level, starting with a single dose (part A) much lower than is expected to cause an effect. Subjects are admitted to a Unit so they can be closely observed for adverse effects and safety tests, blood concentrations of the drug and food and liquid intake and output will be monitored. Subjects are allocated at random (like tossing a coin) to receive Y242 or placebo (dummy). Safety, tolerability and pharmacokinetic data will be summarised and available results considered in deciding dose escalation, with stopping rules designed to enable us to explore the relationship between dose and adverse effect (eg nausea) without causing unacceptable nausea or other symptoms in the volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult males aged 18 to 50 years inclusive with BMI between 23.0 and 30.0 kg/m^2 inclusive;
* Subjects who are healthy as determined by pre study medical history, physical examination and 12 lead ECG;
* Subjects whose clinical laboratory test results are either within the normal range or if outside this range the abnormalities are judged to be not clinically relevant and are acceptable to the Investigator;
* Subjects who are negative for hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) I and II tests at screening;
* Subjects who are negative for drugs of abuse and alcohol tests at screening and admissions;
* Subjects who are non-smokers for at least 3 months preceding screening;
* Subjects who agree to use medically acceptable methods of contraception for at least 3 months after study drug administration;
* Subjects who are able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who do not conform to the above inclusion criteria;
* Subjects who have a clinically relevant history or presence of gastrointestinal (especially associated with vomiting), respiratory, renal, hepatic, haematological, lymphatic, neurological (especially if associated with balance disorders or vomiting e.g. migraine or labyrinthitis), cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders;
* Subjects who have a clinically relevant surgical history;
* Subjects who have a clinically relevant family history;
* Subjects who have a history of relevant atopy;
* Subjects who have a history of relevant drug hypersensitivity;
* Subjects who have a history of alcoholism;
* Subjects who have a history of drug abuse;
* Subjects who have a history of migraine;
* Subjects who consume more than 21 units of alcohol a week (unit = 1 glass of wine (125 mL) = 1 measure of spirits = ½ pint of beer);
* Subjects who have a significant infection or known inflammatory process on screening;
* Subjects who have acute gastrointestinal symptoms at the time of screening or admission (e.g. nausea, vomiting, diarrhoea, heartburn);
* Subjects who have an acute infection such as influenza at the time of screening or admission;
* Subjects who have used prescription drugs within 4 weeks of first dosing;
* Subjects who have used over the counter medication excluding routine vitamins and paracetamol but including megadose (intake of 20 to 600 times the recommended daily dose) vitamin therapy within 7 days of first dosing, unless agreed as not clinically relevant by the Principal Investigator and Sponsor;
* Subjects who have donated blood or blood products within 3 months of Day -2 (admission);
* Subjects who have used any investigational drug in any clinical trial within 3 months of Day -2 (admission);
* Subjects who have received the last dose of investigational drug greater than 3 months ago but who are on extended follow-up;
* Subjects who have previously received Y242;
* Subjects who are vegans or have any dietary restrictions;
* Subjects who cannot communicate reliably with the Investigator;
* Subjects who are unlikely to co-operate with the requirements of the study;
* History or evidence of abnormal eating behaviour, as observed through the Dutch Eating Behaviour (DEBQ) and SCOFF questionnaires at screening.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adult males aged 18 to 50 years inclusive with BMI between 23.0 and 30.0 kg/m^2 inclusive
Enrollment: 68 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bloom DSc, MD FRCP, Study Chair — Imperial College London; John Lambert, MBBS PhD, Principal Investigator — Parexel; Tricia Tan BSc MRCP, MB ChB, Study Director — Imperial College London
Locations (1):
- PAREXEL Early Phase Clinical Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 2mg Y242; 7.5mg Y242; 15mg Y242; 30mg Y242; 60mg Y242; 90mg Y242: Y242 single dose, subcutaneous (Part A)
- 60mg Y242 (B1); 90mg Y242 (B2-B4): Y242 single subcutaneous dose, administered once a week for 5 weeks (Part B)
- Placebo - Part B: 0.9% saline - placebo
Period: Overall Study
Arm/Group | 2mg Y242 | 7.5mg Y242 | 15mg Y242 | 30mg Y242 | 60mg Y242 | 90mg Y242 | Placebo - Part A | 60mg Y242 (B1) | 90mg Y242 (B2-B4) | Placebo - Part B
Started | 3 | 3 | 6 | 6 | 6 | 6 | 10 | 6 | 14 | 8
Completed | 3 | 3 | 6 | 6 | 6 | 6 | 9 | 6 | 9 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2mg Y242 | 7.5mg Y242 | 15mg Y242 | 30mg Y242 | 60mg Y242 | 90mg Y242 | Placebo - Part A | 60mg Y242 (B1) | 90mg Y242 (B2-B4) | Placebo - Part B | Total
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 10 | 6 | 14 | 8 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (2.52) | 39.7 (5.51) | 25.5 (5.79) | 28.7 (9.2) | 31.5 (11.47) | 34.3 (7.5) | 31.3 (6.04) | 35.7 (6.62) | 29.4 (7.1) | 34.6 (6.76) | 31.6 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 6 | 6 | 6 | 6 | 10 | 6 | 14 | 8 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  Black or African American | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 7
  White | 2 | 3 | 4 | 3 | 6 | 5 | 6 | 6 | 9 | 7 | 51
  More than one race | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 3 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Origin: Hispanic Or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 4
  Ethnic Origin: Not Hispanic Or Latino | 3 | 3 | 6 | 5 | 6 | 6 | 8 | 5 | 14 | 8 | 64
Region of Enrollment [Number; unit: participants]
  United Kingdom | 3 | 3 | 6 | 6 | 6 | 6 | 10 | 6 | 14 | 8 | 68
Height (cm) [Mean (Standard Deviation); unit: cm] | 183.3 (8.39) | 174.3 (5.69) | 177.2 (5.71) | 180.8 (9.99) | 177.7 (4.97) | 179.0 (4.29) | 176.5 (6.82) | 174.3 (7.09) | 179.9 (6.32) | 180.9 (6.58) | 178.3 (6.55)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 87.5 (2.893) | 80.27 (7.199) | 84.58 (7.618) | 83.63 (10.723) | 82.52 (11.618) | 83.28 (9.781) | 81.10 (10.363) | 76.18 (7.537) | 84.37 (7.846) | 89.89 (7.906) | 83.5 (9.01)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 26.13 (1.845) | 26.37 (0.929) | 26.88 (1.148) | 25.55 (2.128) | 26.05 (2.595) | 25.93 (2.325) | 25.94 (1.731) | 25.03 (1.462) | 26.07 (1.920) | 27.46 (1.431) | 26.2 (1.84)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment Emergent Adverse Events (TEAEs)
Description: A treatment-emergent AE (TEAE) as defined as an AE that started after administration of IMP; in Part B this was an AE that started after the first dose of IMP. Adverse events with onset prior to dosing were considered as pre-treatment AEs.
Time Frame: Up to 73 days
Population: Summary statistics included number of subjects, arithmetic mean and standard deviation.
Measure: Count of Participants; unit: Participants
Arm/Group | 2mg Y242 | 7.5mg Y242 | 15mg Y242 | 30mg Y242 | 60mg Y242 | 90mg Y242 | Placebo - Part A | 60mg Y242 (B1) | 90mg Y242 (B2-B4) | Placebo - Part B
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 6 | 10 | 6 | 14 | 8
Participants
  Total number of AEs | 0 | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 14 | 7
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs leading to discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Body Weight
Description: Summary of Time-Matched % Change from Baseline in Body Weight (Baseline = Day -1) following multiple dose of Y242 (Part B)
Time Frame: up to 32 day
Population: Part B - Body weight change from baseline (%) following 5 weekly doses of Y242
Measure: Mean (Standard Deviation); unit: Percentage change in Body weight
Arm/Group | 2mg Y242 | 7.5mg Y242 | 15mg Y242 | 30mg Y242 | 60mg Y242 | 90mg Y242 | Placebo - Part A | 60mg Y242 (B1) | 90mg Y242 (B2-B4) | Placebo - Part B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 9 | 8
Percentage change in Body weight |  |  |  |  |  |  |  | -1.2 (1.9) | -1.0 (1.8) | 1.8 (3.4)

ADVERSE EVENTS:
Time Frame: 73 days until final follow up visit
Description: The subjects were queried regularly on all study days using non-leading questions, such as "How do you feel?" In addition, all AEs reported spontaneously during the course of the study were recorded.
Arm/Group | 2mg Y242 | 7.5mg Y242 | 15mg Y242 | 30mg Y242 | 60mg Y242 | 90mg Y242 | Placebo - Part A | 60mg Y242 (B1) | 90mg Y242 (B2-B4) | Placebo - Part B
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/14 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/6 | 0/14 | 0/8
Other Adverse Events (participants affected / at risk) | 0/3 | 3/3 | 6/6 | 6/6 | 6/6 | 6/6 | 6/10 | 6/6 | 14/14 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2mg Y242 (N=3) | 7.5mg Y242 (N=3) | 15mg Y242 (N=6) | 30mg Y242 (N=6) | 60mg Y242 (N=6) | 90mg Y242 (N=6) | Placebo - Part A (N=10) | 60mg Y242 (B1) (N=6) | 90mg Y242 (B2-B4) (N=14) | Placebo - Part B (N=8)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 5 (5) | 4 (4) | 0 (0) | 4 (12) | 14 (39) | 1 (1)
Tooth Ache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza-like Illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site Discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Induration (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Reaction (General disorders) | 0 (0) | 3 (4) | 5 (7) | 5 (7) | 6 (6) | 6 (7) | 1 (1) | 6 (29) | 14 (58) | 1 (1)
Gastoenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Catheter Site Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 5 (10) | 3 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal Hypoaestesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling of Body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes